CLINICAL TRIAL: NCT04689243
Title: Clinical Study of Low Concentration ALA-PDT in Treatment of Skin Ulcer
Brief Title: Low Concentration ALA-PDT in Treatment of Skin Ulcer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yujie Mao, principal investigator, Sichuan Provincial People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2018QN02
Record Dates: First submitted 2020-12-23; First posted 2020-12-30 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Skin Ulcer; Photodynamic Therapy
MeSH Terms: conditions — Skin Ulcer | interventions — Red Light

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ALA-PDT (Experimental)
  Interventions: Procedure: ALA-PDT
- red light (Other)
  Interventions: Procedure: red light

INTERVENTIONS:
Procedure: ALA-PDT — Low concentration ALA-PDT, 3 times a week.
  Arms: ALA-PDT
Procedure: red light — red light, 3 times a week.
  Arms: red light

SUMMARY:
Skin ulcer is a common disease with complicated etiopathogenes, which makes it hard to be cured. It has been reported that photodynamic therapy (PDT) can be used to treat skin ulcers which were caused by different diseases. However, PDT is an expensive treatment and patients always experience obvious pain during or after the treatment, which hinders the application of PDT in skin ulcer. Our previous study found that PDT using a low concentration of 5-Aminolevulinic acid (ALA) could promote the healing of skin ulcer without obvious adverse reactions, which suggests us that low concentration ALA-PDT might be an efficient and cost effective treatment in skin ulcer. To further investigate the use of low concentration ALA-PDT in skin ulcer, we plan to recruit patients with skin ulcers caused by different diseases, and divide these patients into different groups according to their causes of disease, and then treat them using low concentration ALA-PDT to observe the healing process of skin ulcer. This study could further optimize and promote the use of low concentration ALA-PDT in skin ulcer.

ELIGIBILITY:
Inclusion Criteria:

* chronic skin wounds that involved the dermis and did not heal in three months or did not exhibit a tendency toward healing

Exclusion Criteria:

* allergies to photosensitizers and their solvents, serious medical illnesses, such as severe heart disease, severe liver or kidney dysfunction, systemic infection or any concomitant infection that would require treatment with an additional antimicrobial agent, the use of topical or systemic antibiotics within one month prior to treatment. Pregnant or lactating women were also excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-12-26 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
ulcer area size | Change from Baseline ulcer area size at 24 hours after the last treatment.
  The ulcer area size was measured

SECONDARY OUTCOMES:
total bacterial load | Change from Baseline total bacterial load at 24 hours after the last treatment.
  Levels of total bacteria were tested

CONTACTS AND LOCATIONS:
Locations (1):
- Sichuan Provincial People's Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Undecided